CLINICAL TRIAL: NCT05326971
Title: The Effect of Tenofovir Disoproxil Fumarate (TDF) Versus Tenofovir Alafenamide (TAF) on Proximal Small Intestine - a Potential Mechanism to Explain Opposing Effects on Body Weight
Brief Title: The Effect Tenofovir Disoproxil Fumarate (TDF) and Tenofovir Alafenamide (TAF) on Small Intestine Gut Wall
Acronym: TENENTOX
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jussi Sutinen (Other)
Collaborators: Helsinki University Central Hospital (Other); University of Helsinki (Other)
Responsible Party: Sponsor-Investigator, Jussi Sutinen, Infectious Disease Consultant, Helsinki University Central Hospital
Organization: Helsinki University Central Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1/2022
Record Dates: First submitted 2022-03-27; First posted 2022-04-14 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: HIV Infections; Weight Gain
Keywords: tenofovir disoproxil fumarate; tenofovir alafenamide; gastroscopy; mitochondria
MeSH Terms: conditions — HIV Infections; Weight Gain | interventions — Gastroscopy

STUDY DESIGN:
Intervention Model Description: A cross sectional study recruiting participants with their own regular home medication.
Who Masked: Outcomes Assessor
Masking Description: Pathologist and mitochondrial researchers performing biopsy studies are blinded for the study groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tenofovir disoproxil TDF (Experimental): Participants who have used TDF as part of their stable antiretroviral regimen for at least past six months.
  Interventions: Procedure: gastroscopy
- Tenofovir alafenamide (TAF) (Active Comparator): Participants who have used TAF as part of their stable antiretroviral regimen for at least past six months.
  Interventions: Procedure: gastroscopy

INTERVENTIONS:
Procedure: gastroscopy — Gastroscopy to evaluate the effect of long term exposure of TDF or TAF on enterocytes

SUMMARY:
Several studies among people living with HIV (PLWH) have shown more weight gain with tenofovir alafenamide (TAF) than with tenofovir disoproxil fumarate (TDF). This difference could be due to weight increasing effect of TAF and / or weight decreasing effect of TDF.

When TDF is ingested, it gets absorbed in the beginning of the small intestine. TDF is processed into free tenofovir (TFV) within the enterocytes, whereas TAF is not. The effect of TFV on enterocytes is not known, but in kidney tubular cells TFV seems to damage mitochondria and that seems lead to TDF-associated kidney toxicity.

In the present cross sectional study the investigators hypothesize that TDF but not TAF causes damage in the small intestine gut wall and that may lead to poorer absorption of nutrients and opposing effects on body weigh.

Twelve stable PLWH who have been treated with TDF for at least past 6 months and 12 PLWH who have similarly been treated with TAF for at least past 6 months will be recruited. The participants will have a gastroscopy done with biopsies taken from the small intestine. These biopsies will be examined for mitochondrial damage and other potential pathological findings. In addition, blood concentrations of several nutrients absorbed from the same part of the small intestine as TDF and blood concentrations of some markers of intestinal damage will be measured.

DETAILED DESCRIPTION:
Integrase inhibitors (INSTI) and tenofovir alafenamide (TAF) have been associated with increased weight gain in several randomized studies among people living with HIV (PLWH). In most of these studies, the control group received tenofovir disoproxil (TDF) which raises the question whether the difference in weight change is due to weight increasing effect of INSTI/TAF or weight decreasing effect of TDF.

When ingested, TDF is prone to chemical and enzymatic hydrolysis by intestinal esterases once pH rises above 3. Therefore, it has a narrow time window to be absorbed as an intact prodrug from the proximal small intestine, also the site of absorption of considerable proportion of lipids, lipid-soluble vitamins, folates, calcium, phosphate, iron, and other micronutrients.

TDF is metabolized within enterocytes in a two-step process of ester group cleavage into free phosphonate tenofovir (TFV). Neither TDF nor the monoester intermediate are detected in systemic circulation, indicating complete presystemic metabolism. The consequences of free TFV within enterocytes are not known, but TFV is cytotoxic in renal tubular cells.

TAF is more resistant than TDF to enzymatic hydrolysis. Due to the smaller amount of ingested prodrug and based on PK studies, it is suggested that ingestion of TAF leads to much smaller - if any - intracellular concentration of TFV within enterocytes than that of TDF.

Mechanisms behind these clinical effects of TDF are not known. The investigators hypothesize these effects are mediated by reduced absorptive function of the proximal small intestine caused by intracellular accumulation of free TFV within enterocytes, a parallel mechanism to TFV-induced toxicity in proximal tubular cells.

This is a cross-sectional study comprising 24 adult PLW on stable antiretroviral therapy containing either TDF (n=12) or TAF (n=12) for at least the past six months. All participants will have a gastroduodenoscopy with biopsies from proximal and distal duodenum. Blood concentrations of nutrients absorbed from the proximal small intestine and related substances will be measured, as well as circulating markers of intestinal damage and function.

The primary objective is to compare pathology findings including mitochondrial studies in duodenal biopsies of PLWH receiving either TDF or TAF. The secondary objectives are to compare the effects of TDF versus TAF on absorption of selected nutrients absorbed from proximal duodenum and circulating markers of intestinal damage and function and microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 year;
* HIV-positive on a stable ART including either TDF or TAF for > 6 months
* HIV viral load < 200 copies for ≥ 6 months.

Exclusion Criteria:

* Known or suspected enteropathies (celiac disease, inflammatory bowel disease)
* Use of any of the following during the previous month: calcium, folic acid, iron, vitamin A, B, E supplements
* Pregnancy.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-01-19 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Mitochondrial respiratory chain function in situ | Baseline
  Cytochrome C Oxidase / Succinate Dehydrogenase (COX/SDH) activity analysis from cryosections
Histopathology of duodenal biopsies | Baseline
  Modified Marsh Classification

SECONDARY OUTCOMES:
Fasting plasma lipid concentrations | Baseline
  total, LDL and HDL cholesterol and triglycerides (all values in mmol/L)
Fasting plasma calcium concentration (fP-Ca-ion) | Baseline
  mmol/l
Fasting serum folate concentration (fS-folate) | Baseline
  nmol/l
Fasting plasma iron concentration (fP-Fe) | Baseline
  umol/l
Fasting serum beta carotene concentration (fS-beta carotene) | Baseline
  nmol/l
Fasting blood thiamine concentration (fB-B1vit) | Baseline
  nmol/l
Fasting serum intestinal fatty acid binding protein (fS-IFABP2) | Baseline
  ng/mL

CONTACTS AND LOCATIONS:
Overall Officials: Jussi Sutinen, Principal Investigator — Helsinki University Hospital Infectious Disease Clinic
Locations (1):
- Infectious Disease Clinic, Helsinki University Hospital, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kauppinen KJ, Aho I, Sjoblom N, Tynninen O, Suomalainen A, Schwab U, Zhao F, Arkkila P, Sutinen J. Effect of 2 Forms of Tenofovir on Duodenal Enterocytes-A Hypothesis for Different Effect of Tenofovir Disoproxil Fumarate and Tenofovir Alafenamide on Body Weight and Plasma Lipids. Clin Infect Dis. 2025 Feb 24;80(2):381-388. doi: 10.1093/cid/ciae374. PMID 39039812